CLINICAL TRIAL: NCT04332081
Title: Open Label Single-Center Study of Emergency Hyperbaric Oxygen for Respiratory Distress in Patients With COVID-19
Brief Title: Hyperbaric Oxygen for COVID-19 Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The IRB has determined that the design of this trial should be changed to a randomized controlled trial. A new record will be created for the redesigned study.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-00399
Record Dates: First submitted 2020-03-30; First posted 2020-04-02 (Actual); Results first posted 2021-06-22 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: prospective pilot cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Hyperbaric oxygen therapy (HBOT) (Experimental)
  Interventions: Device: hyperbaric oxygen therapy (HBOT)
- Standard of Care (No Intervention)

INTERVENTIONS:
Device: hyperbaric oxygen therapy (HBOT) — The patient will receive 90 minutes of hyperbaric oxygen at 2.0 ATA with or without airbreaks per the hyperbaric physician. Upon completion of the treatment the patient will then return to the medial unit and continue all standard of care. Additional treatments (up to 5) can be given if warranted and agreed upon by the patient and all members of the team caring for the patient.
  Arms: Hyperbaric oxygen therapy (HBOT)

SUMMARY:
Hyperbaric oxygen therapy (HBOT) treatment will be provided to patients as an adjunct to standard therapy for a cohort of 40 COVID19-positive patients with respiratory distress at NYU Winthrop Hospital. All patients prior to the clinical application of HBOT will be evaluated by the primary care team and hyperbaric physician. After the intervention portion of this study, a chart review will be performed to compare the outcomes of intervention patients versus patients who received standard of care.

DETAILED DESCRIPTION:
This is a single center prospective pilot cohort study to evaluate the safety and efficacy of hyperbaric oxygen therapy (HBOT) as an emergency investigational device for treating patients with a novel coronavirus, disease, COVID-19. Patients that meet inclusion criteria will be consented by the hyperbaric physician. They will then be transported from the ED or other unit to the hyperbaric unit maintaining airborne precautions based on the most current hospital protocol. All study personnel will have proper PPE at all times. The patient will then be placed into the monoplace chamber and when the chamber door is closed the patient will remove any respiratory filter/mask that was placed. The patient will receive 90 minutes of hyperbaric oxygen at 2.0 ATA with or without airbreaks per the hyperbaric physician. Upon completion of the treatment the patient will then return to the medical unit and continue all standard of care. Additional treatments (up to 5) can be given if warranted and agreed upon by the patient and all members of the team caring for the patient. After the intervention portion of this study, a chart review will be performed to compare the outcomes of intervention patients versus patients who received standard of care.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Male or female, age > 18 years
2. Positive COVID 19 test
3. Respiratory compromise defined by SpO2 <93%
4. Ability to sign informed consent

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Pregnancy
2. Untreated Pneumothorax

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-05-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- NYU Winthrop Hospital, Mineola, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be made available immediately following publication, upon reasonable request by an investigator who proposes to use the data.
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication. No end date.
Access Criteria: Requests should be directed to David.Lee@nyulangone.org and Scott.Gorenstein@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: No HBOT
Period: Overall Study
Arm/Group | Hyperbaric Oxygen Therapy (HBOT) | Standard of Care
Started | 20 | 60
Completed | 20 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hyperbaric Oxygen Therapy (HBOT) | Standard of Care | Total
Number analyzed (Participants) | 20 | 60 | 80
Age, Continuous [Mean (Full Range); unit: years] | 58 [30 to 79] | 62 [24 to 80] | 60 [24 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 18 | 55 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 20 | 60 | 80
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 6 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 10 | 13
  White | 7 | 16 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 28 | 37
Region of Enrollment [Number; unit: participants]
  United States | 20 | 60 | 80

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Time Frame: through study completion; an average of 50 days
Measure: Number; unit: % of participants
Arm/Group | Hyperbaric Oxygen Therapy (HBOT) | Standard of Care
Number analyzed (Participants) | 20 | 60
% of participants | 10 | 22

2. Secondary Outcome: Need for Mechanical Ventilation
Time Frame: through study completion; an average of 50 days
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Oxygen Therapy (HBOT) | Standard of Care
Number analyzed (Participants) | 20 | 60
Participants | 2 | 18

ADVERSE EVENTS:
Time Frame: through study completion; an average of 50 days
Arm/Group | Hyperbaric Oxygen Therapy (HBOT) | Standard of Care
All-Cause Mortality (participants affected / at risk) | 2/20 | 13/60
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/60
Other Adverse Events (participants affected / at risk) | 0/20 | 0/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hyperbaric Oxygen Therapy (HBOT) (N=20) | Standard of Care (N=60)
Hypoxic Arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/81/NCT04332081/Prot_SAP_000.pdf